CLINICAL TRIAL: NCT03721198
Title: Resin-modified Glass Ionomer Varnish Versus Acidulated Phosphorus Fluoride Gel in Prevention of White Spot Lesions During Comprehensive Orthodontic Treatment: (Split Mouth Randomized Clinical Trial)(A Comparative Study)
Brief Title: RMGI Varnish Versus APF Gel in Prevention of White Spot Lesions During Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohamed zidan (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Mohamed zidan, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMGI Varnish-WSL prevention
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: White Spot Lesion of Tooth

STUDY DESIGN:
Intervention Model Description: split mouth technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acidulated phosphorous flouride (Active Comparator): Acidulated phosphorous flouride used once at the first of the study
  Interventions: Combination Product: Acidulated phosphorous flouride
- Resin modified glass ionomer varnish (Experimental): Resin modified glass ionomer varnish (CLINPRO XT ) is used once at the first of the study only
  Interventions: Other: Resin modified glass ionomer varnish

INTERVENTIONS:
Combination Product: Acidulated phosphorous flouride — Acidulated phosphorous flouride is used to prevent white spot lesions
  Other Names: APF
  Arms: Acidulated phosphorous flouride
Other: Resin modified glass ionomer varnish — Resin modified glass ionomer varnish is used to prevent white spot lesions
  Other Names: CLINPRO XT
  Arms: Resin modified glass ionomer varnish

SUMMARY:
evaluate the effect of a single application of Clinpro XT varnish on enamel demineralization adjacent to orthodontic brackets during fixed orthodontic treatment in comparison with acidulated phosphorus fluoride gel.

this study is to assess the durability of the results obtained from both materials (Clinpro XT Varnish- APF Gel) this study is to determine the degree of

patients' satisfaction after the use of both materials (Clinpro XT Varnish -

APF Gel)

DETAILED DESCRIPTION:
This clinical study will be held in the orthodontic clinic, Faculty of dentistry, Cairo University, Egypt Principal investigator (MZ) will select and examine the patients according to the inclusion criteria.

Tooth preparation procedure:

Excessive saliva in Upper six anterior teeth will be removed by cotton rolls or by using an air syringe without excessive drying. Principal investigator (MZ) will take a photograph for each tooth using A Digital DSLR camera (canon 700d with lens 100 macro 2.8) and this photograph is T0(before application of the gel)

Intervention and comparator:

1. Bonding procedure before application of intervention and comparator

   Upper six anterior teeth will be cleaned with pumice, rinsed and dried thoroughly. The area where the bracket is to be placed will be etched with a 37% orthophosphoric acid gel for 15 seconds and then rinsed with water. After rinsing, the enamel surface will be dried with compressed moisture and oil free air. A layer of primer will be applied to the tooth and bracket mesh. Adhesive paste will be applied to the base of the bracket and pressed firmly onto the tooth surface. Excess adhesive will be removed, and the adhesive light cured for 20 seconds.
2. Preparation of clinpro XT (intervention)

   In upper right anterior teeth, the polished tooth surface is etched using 37% orthophosphoric acid gel. applied for 15 seconds over the labial enamel surface extending from gingival surface of the bracket to the free gingival margin. Then, the surface is rinsed thoroughly by water spray and dried with compressed moisture and oil free air to remove the etchant. The paste and liquid components of the varnish are mixed on a paper pad for 10-15 seconds by a small plastic spatula. When the mix material appears glossy and smooth in consistency, it is applied as a thin layer over the etched enamel surface by a ball applicator. Care should be taken to avoid prolonged contact of uncured material with soft tissues.

   If accidental contact occurred, the material is immediately wiped off with wet cotton roll. Then, the varnish is light cured with the visible light-curing unit for 20 s.Oral hygiene instruction will be given to the patient e.g. tooth brushing twice a day with fluoride toothpaste.

   A photograph will be taken for the labial surface of each upper right anterior tooth using the same camera by the outcome assessor (MS) after 3 months (T1) and 6 months (T2) of orthodontic treatment.
3. Preparation of Acidulated Phosphorus Fluoride (Comparator):

Acidulated Phosphorus Fluoride gel will be applied directly over the labial enamel surface extending from gingival surface of the bracket to the free gingival margin using a small brush/swab to spread the gel over the surface. The gel will be left in place for four minutes then washed. Patients will be instructed not to rinse, eat, drink or smoke for the next 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicating for fixed orthodontic treatment with healthy gingival and periodontal condition

Exclusion Criteria:

1. Presence of enamel hypoplasia or dental fluorosis.
2. Presence of tetracycline pigmentation.
3. Periodontal pocketing of 3mm or greater.
4. Presence of carious cavities.
5. Smokers.
6. Allergy to fluoride gel being used in study.
7. Patient that have systemic disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Colour change | 6 months
  Colour change using spectrophotometer

SECONDARY OUTCOMES:
Colour stability | 6 months
  Colour stability using spectrophotometer

OTHER OUTCOMES:
Patient satisfaction: VAS APF Gel) | 6 months
  Patient satisfaction using visual analogue scale A scale to assess the patient satisfaction A scale from 0 to 10 10 means fully satisfied by the results 0 means unsatisfied by the result

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Saied, Study Chair — orthodontic department

IPD SHARING:
Plan to Share IPD: Undecided